CLINICAL TRIAL: NCT04042298
Title: Microvascular Function in Patients Undergoing 5-Fluorouracil Chemotherapy
Status: Completed | Type: Observational
Sponsor: Kansas State University (Other)
Responsible Party: Principal Investigator, Carl Ade, M.S., Ph.D., Assistant Professor, Kansas State University
Other Study IDs: Pro9646
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Gastrointestinal Cancer; Head and Neck Cancer; Breast Cancer; Chemotherapy Effect; 5-Fluorouracil Toxicity
MeSH Terms: conditions — Gastrointestinal Neoplasms; Head and Neck Neoplasms; Breast Neoplasms | interventions — Arterial Pressure; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples (5-7 mL) from the antecubital vein or a vein in the back of the hand will be taken via venipuncure by a nurse or a certified phlebotomist at the beginning of the experimental visit. These blood samples will be analyzed for the presence of reactive oxygen species and inflammatory markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- 5-FU Chemotherapy (Experimental): Comprised of newly diagnosed cancer patients 21 years or older who have received 5-FU chemotherapy within the past 30 days or are scheduled to receive 5-FU chemotherapy.
  Interventions: Other: Arterial blood pressure; Other: Skin microcirculatory blood flow; Other: Brachial artery blood flow; Other: Venous blood draw
- Non-5-FU Chemotherapy (Sub-Control): Comprised of newly diagnosed cancer patients 21 years or older who have received chemotherapy other than 5-FU within the past 30 days or are scheduled to receive chemotherapy other than 5-FU.
  Interventions: Other: Arterial blood pressure; Other: Skin microcirculatory blood flow; Other: Brachial artery blood flow; Other: Venous blood draw
- Age/Sex matched Control (Control): Age, biological sex, and prior health history (excluding cancer diagnosis) matched control for cancer patients
  Interventions: Other: Arterial blood pressure; Other: Skin microcirculatory blood flow; Other: Brachial artery blood flow; Other: Venous blood draw
- 5-FU Chemotherapy Cancer Survivor (Survivor): Cancer survivors who have not received cancer therapy during the past year but previously received 5-Fluorouracil chemotherapy.
  Interventions: Other: Arterial blood pressure; Other: Skin microcirculatory blood flow; Other: Brachial artery blood flow; Other: Venous blood draw

INTERVENTIONS:
Other: Arterial blood pressure — Measured using an automated non-invasive finger cuff that obtains beat-by-beat blood pressure measurements via finger photoplesmography. Briefly, changes in artery diameter are detected through infrared light in the finger cuff. (Finometer Pro, FMS, The Netherlands).
Other: Skin microcirculatory blood flow — Assessed non-invasively in the forearm skin via Laser Doppler flowmetry in response to locally delivered acetylcholine and norepinepherine or phenylepherine via iontophoresis.
Other: Brachial artery blood flow — A GE Ultrasound System will be used to non-invasively assess brachial artery blood flow prior to and following a standard flow mediated dilation protocol.
Other: Venous blood draw — A venous blood sample from the antecubital vein or a vein in the back of the hand will be taken via venipuncure by a nurse or a certified phlebotomist at the beginning of the experimental visit. These blood samples will be analyzed for the presence of reactive oxygen species and inflammatory markers.

SUMMARY:
The primary aim of this study is to investigate potential differences in vascular function between patients receiving 5-Fluorouracil (5-FU) chemotherapy, patients receiving chemotherapies other than 5-FU, cancer survivors who were treated with 5-FU, and an age and sex matched control. 5-FU is the third most commonly administered chemotherapeutic agent and its use is associated with the second most occurrences of cardiotoxicity. Despite the known cardiotoxic effects of 5-FU, it's effects on the human vasculature are not well understood.

To achieve the goals of this project Laser Doppler flowmetry (LDF) will be used to assess blood flow within the skin microcirculation of the forearm in cancer patients who have received 5-Fluoruracil within the past 30 days (Experimental Group), cancer patients receiving radiotherapy and/or chemotherapy other than 5-Fluorouracil, and an age and sex matched control (Control Group). LDF utilizes a small (~3 cm) non-invasive sensor placed on the skin. The sensor shines light into the skin, and upon contact with red blood cells (RBCs), the light is reflected and scattered. This information is used to evaluate microvascular blood flow and has previously been used in clinical populations.

DETAILED DESCRIPTION:
Although cancer continues to be one of the leading causes of death each year, advancements in cancer treatments and detection have improved patient prognosis across a large number of cancer types. This trend of improved survival rates has made apparent the significant risk of chemotherapy on the cardiovascular system in such a way that cardiotoxicity has become a prime concern in cancer survivors. Indeed, cardiotoxic events have been related to numerous chemotherapy types, including the commonly used 5-Fluorouracil (5-FU). 5-FU is the third most commonly administered form of chemotherapy used in the treatment of solid malignancies. Despite undeniable effectiveness in treating cancer, administration of 5-FU is associated with the second highest incidence of cardiotoxicity out of all chemotherapeutic agents.

Such cardiotoxic manifestations typically appear in the form of chest pain, angina during rest and/or exertion, and acute coronary syndromes, however, other events such as arrythmias, myocarditis, pericarditis, heart failure, or even death have been reported following 5-FU administration. While multiple mechanisms are believed to lead to 5-FU cardiotoxicity, the effects 5-FU has on the vasculature seem to be of particular importance. Initial findings suggest these drugs have a direct toxic effect on the vascular endothelium and smooth muscle, likely through increases in reactive oxygen species (ROS). ROS are known to adversely affect endothelium independent and dependent factors which influence vascular tone. Along with increased ROS, decreases in antioxidant capacity following 5-FU therapy lead to increased vasospasms and altered vasodilator/constrictor responses. Indeed, both coronary artery vasospasms and brachial artery vasoconstriction have been found to occur in some groups directly after injection of 5-FU.

Although the primary signaling pathways for 5-FU induced cardiotoxicity are well documented, many of these studies have been conducted in animal models. Previous work has demonstrated substantial vascular dysfunction in current cancer patients undergoing adjuvant systematic chemotherapy when compared to healthy controls, however, alike investigations specifically focused on vascular dysfunction in patients receiving 5-FU have yet to be conducted. To investigate such mechanisms, microvascular reactivity will be measured with laser Doppler flowmetry combined with iontophoresis of acetylcholine in cancer patients currently undergoing treatment with 5-Fluorouracil, patients receiving chemotherapy treatments other than 5-Fluorouracil, cancer survivors previously treated with 5-Fluorouracil, and age and sex matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study
* (Group 1) Current cancer treatment includes 5-FU
* (Group 2) Current cancer treatment does not include 5-FU
* (Group 3) Cancer survivor previously treated with 5-FU but has not received cancer treatment in the year proceeding enrollment.
* (Group 4) Age, sex, and health matched (excluding cancer) control for Group 1

Exclusion Criteria:

* (Groups 1, 2, and 4) Have received cancer treatment outside of the past year
* Not met above criteria
* Pregnant, breastfeeding, or planning to become pregnant
* Unable to provide informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed cancer patients who have received (or are scheduled to receive) 5-FU chemotherapy within the past 30 days (n=26) will enter the study soon after initiation of treatment. Newly diagnosed cancer patients receiving cancer treatment other than 5-FU (n=26; chemotherapy, radiotherapy, etc.) will enter into the study soon after initiation of treatment. Cancer survivors (n=26) who have previously received 5-FU but not within the year proceeding enrollment will be entered into the study. Age, sex, and health (n=26; excluding cancer) matched controls will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Cutaneous (skin) blood flow (%) following administration of vasoactive substances | 1 day
  Measured once in each group following administration of vasodilatory (Acetylcholine) and vasoconstrictive (Norepinepherine or Phenylephrine) substances.
Brachial artery flow mediated dilation (FMD) | 1 day
  Measured once in each group

SECONDARY OUTCOMES:
Arterial blood pressure | 1 day
  Systolic, diastolic, and mean arterial pressure will be measured continuously over the course of the visit for each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Lafene Health Center, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yeh ET, Bickford CL. Cardiovascular complications of cancer therapy: incidence, pathogenesis, diagnosis, and management. J Am Coll Cardiol. 2009 Jun 16;53(24):2231-47. doi: 10.1016/j.jacc.2009.02.050. PMID 19520246
- [Background] Sara JD, Kaur J, Khodadadi R, Rehman M, Lobo R, Chakrabarti S, Herrmann J, Lerman A, Grothey A. 5-fluorouracil and cardiotoxicity: a review. Ther Adv Med Oncol. 2018 Jun 18;10:1758835918780140. doi: 10.1177/1758835918780140. eCollection 2018. PMID 29977352
- [Background] Taniyama Y, Griendling KK. Reactive oxygen species in the vasculature: molecular and cellular mechanisms. Hypertension. 2003 Dec;42(6):1075-81. doi: 10.1161/01.HYP.0000100443.09293.4F. Epub 2003 Oct 27. PMID 14581295
- [Background] Polk A, Vistisen K, Vaage-Nilsen M, Nielsen DL. A systematic review of the pathophysiology of 5-fluorouracil-induced cardiotoxicity. BMC Pharmacol Toxicol. 2014 Sep 4;15:47. doi: 10.1186/2050-6511-15-47. PMID 25186061
- [Background] Luwaert RJ, Descamps O, Majois F, Chaudron JM, Beauduin M. Coronary artery spasm induced by 5-fluorouracil. Eur Heart J. 1991 Mar;12(3):468-70. doi: 10.1093/oxfordjournals.eurheartj.a059919. PMID 2040332
- [Background] Sudhoff T, Enderle MD, Pahlke M, Petz C, Teschendorf C, Graeven U, Schmiegel W. 5-Fluorouracil induces arterial vasocontractions. Ann Oncol. 2004 Apr;15(4):661-4. doi: 10.1093/annonc/mdh150. PMID 15033676
- [Background] Sutterfield SL, Caldwell JT, Post HK, Lovoy GM, Banister HR, Ade CJ. Lower cutaneous microvascular reactivity in adult cancer patients receiving chemotherapy. J Appl Physiol (1985). 2018 Oct 1;125(4):1141-1149. doi: 10.1152/japplphysiol.00394.2018. Epub 2018 Aug 9. PMID 30091663